CLINICAL TRIAL: NCT06823180
Title: Clinical Effect of Hydromorphone Hydrochloride Epidural Preemptive Analgesia on Postoperative Pain After Cesarean Section
Brief Title: Hydromorphone Hydrochloride Epidural Preemptive Analgesia for Postoperative Pain After Cesarean Section
Acronym: HHEPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Liquan Liang (Other)
Responsible Party: Sponsor-Investigator, Liquan Liang, Doctor of Medicine, Jiangxi Provincial People's Hopital
Organization: Jiangxi Provincial People's Hopital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024-128IITFS
Record Dates: First submitted 2025-01-22; First posted 2025-02-12 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Post-surgical Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Hydromorphone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose of hydromorphone hydrochloride was given to the drug group (Experimental): 15min before the end of the operation, 0.1mg hydromorphone hydrochloride was injected epidural into the low-dose group for preemptive analgesia.
  Interventions: Drug: Hydromorphone hydrochloride low dose
- High dose of hydromorphone hydrochloride was given to the drug group (Experimental): 15min before the end of the operation, 0.3mg hydromorphone hydrochloride was injected epidural into the high dose group for preemptive analgesia.
  Interventions: Drug: Hydromorphone hydrochloride high dose
- control group (Placebo Comparator): 15min before the end of the operation, the control group was simply given equal dose 0.9% sodium chloride injection.
  Interventions: Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: Hydromorphone hydrochloride low dose — 15min before the end of the operation, 0.1mg hydromorphone hydrochloride was injected into the epidural space in the low-dose group for preemptive analgesia.
  Arms: Low dose of hydromorphone hydrochloride was given to the drug group
Drug: Hydromorphone hydrochloride high dose — 15min before the end of the operation, 0.3mg hydromorphone hydrochloride was injected into the epidural space in the high-dose group for preemptive analgesia.
  Arms: High dose of hydromorphone hydrochloride was given to the drug group
Drug: 0.9% sodium chloride — 15min before the end of the operation, 0.9% sodium chloride injection was given in the control group.
  Arms: control group

SUMMARY:
Acute pain often occurs after cesarean section, which can lead to stress and inflammatory response in the body, which will not only affect the postpartum recovery speed of the puerpera, but also inhibit the secretion of prolactin to a certain extent and reduce the secretion of milk. Epidural anesthesia is a common anesthesia method for cesarean section, which has the advantages of easy operation and little influence on the fetus. Preemptive analgesia can effectively block the transmission of harmful stimuli and reduce the degree of pain after cesarean section. Hydromorphone hydrochloride is a derivative of morphine, which has the advantages of rapid onset and good analgesic effect, and has been widely used in clinic. However, it is not clear whether epidural injection of hydromorphone hydrochloride for preanalgesia can bring clinical benefits to puerpera, and the optimal dose of hydromorphone hydrochloride for cesarean section is also unclear.

The parturient women who met the inclusion criteria were randomly divided into 3 groups: control group, hydromorphone hydrochloride low-dose administration group and hydromorphone hydrochloride high-dose administration group. All women received epidural combined subarachnoid anesthesia. 15min before the end of the operation, the low-dose hydromorphone hydrochloride group was injected with 0.1mg hydromorphone hydrochloride in the epidural space, the high-dose hydromorphone hydrochloride group was injected with 0.3mg hydromorphone hydrochloride in the epidural space, and the control group was injected with 0.9% sodium chloride injection. Post-obstetric visual analogue scale (VAS) was followed up to record PCA compression times, gastrointestinal peristalsis recovery time, getting out of bed time, lactation time, and related adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Parturients with indications for cesarean section;
* American Association of Anesthesiologists (ASA) Grade I - II;
* No history of sedative drugs or opioid abuse;
* Volunteer to join the study

Exclusion Criteria:

* People with coagulation disorders;
* preoperative use of analgesia, non-steroidal drugs;
* Abnormal liver and kidney function;
* Postoperative drainage is urgently needed.

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Our study focused on women who were expecting to give birth, so we included only women
Enrollment: 105 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
VAS score | 24 hours after surgery
  VAS score was used to evaluate the pain in each period after obstetric surgery. A strip marked with a scale of 0-10 was taken, where 0 indicated no pain, the pain degree increased with the increase of the score, and 10 indicated the most pain. The mothers chose the score matching their own pain degree. Mild pain: 0<VAS<4 ; Moderate pain :4 ≤VAS< 7; Severe pain :7 ≤VAS<9; Extreme pain: VAS≥9.

SECONDARY OUTCOMES:
The number of PCA compressions after surgery | 48 hours after surgery
Satisfaction evaluation | Before discharge
  Patients' satisfaction was assessed by HCAHPS survey. The survey was designed to assess patient inpatient experience, including nurse care, physician communication, hospital environment, hospital experience, discharge information provision, and overall hospital evaluation.
Gastrointestinal peristalsis recovery time | 72 hours after surgery
  The recovery time of bowel sound, anal exhaust and defecation were recorded.
The time it takes to get out of bed for the first time after surgery | 96 hours after surgery
The time between the end of surgery and lactation | 72 hours after surgery
Postoperative nausea and vomiting（PONV） | 72 hours after surgery
  PONV rating standards of WHO are adopted. Specifically: Grade I is no nausea, vomiting; Grade II was mild nausea, abdominal discomfort, but no vomiting; Grade III is nausea and vomiting, but there is no content spit out; Grade IV is severe vomiting, with vomiting of stomach contents and requiring medical control.
pruritus | 72 hours after surgery
  The numeric rating scale (NRS) was used to evaluate the degree of postoperative pruritus. Itching is numerically graded on the NRS scale, with 0 indicating no itching and 10 indicating the most severe itching. The degree of itching increased with the increase of the score. Mild pruritus :0<NRS<4 ; Moderate pruritus :4 ≤NRS< 7; Severe pruritus :7 ≤NRS<9; Extreme pruritus :NRS≥9.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Provincial People's Hospital, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No